CLINICAL TRIAL: NCT04113330
Title: Surveillance of Suspected Dengue Cases for Access to Care for Subjects Identified as Seronegative or Undetermined at Baseline and Who Received CYD Dengue Vaccine in CYD15, CYD13, CYD29, CYD64, CYD65 Trials in Colombia
Brief Title: Surveillance of Suspected Dengue Cases for Access to Care for Subjects Identified as Seronegative or Undetermined Before Receiving CYD Dengue Vaccine in Previous Clinical Studies in Colombia
Acronym: CYD00082
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: CYD00082; U1111-1215-0183 (Registry Identifier: ICTRP)
Record Dates: First submitted 2019-09-26; First posted 2019-10-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Participant vaccinated with CYD Dengue Vaccine and classified as seronegative or undetermined at baseline in previous dengue studies in Colombia

SUMMARY:
The primary objective of the study is to identify any suspected dengue case in subjects that received at least one dose of the CYD dengue vaccine who were classified as seronegative or undetermined at baseline (according to PRNT50 at baseline, or anti-non-structural protein 1 [NS1] test Post-dose 3) in the Colombian study sites of CYD15, CYD13, CYD29, CYD64, CYD65 trials in order to allow appropriate access to care until the completion of 10 years after the last CYD Dengue Vaccine received by each participant

DETAILED DESCRIPTION:
The planned duration of each participant's participation in the study will vary according to the date when they received their last CYD Dengue Vaccine. The surveillance will last during 10 year after the last CYD dengue vaccination of included participants

ELIGIBILITY:
Inclusion Criteria:

* Participants classified as seronegative or undetermined at baseline (by PRNT50 at baseline or anti-NS1 test Post-dose 3) that had received at least one dose of the tetravalent CYD dengue vaccine in the clinical sites of CYD15, CYD13, CYD29, CYD64, or CYD65 studies in Colombia
* Informed consent form or Assent form has been signed and dated by the participant (based on local regulations), and/or informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations)
* Participant (or participant and parent[s] or another legally acceptable representative) is (are) able to comply with all study procedures

Exclusion criteria:

* Participants that were withdrawn from the CYD15, CYD13, CYD29, CYD64, or CYD65 study in Colombia study due to "lost to follow-up" and despite various attempts, were not possible to be contacted
* Participants that cannot be contacted after 3 phone calls, SMS, one home visit and written contact letter/email/WhatsApp

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participant vaccinated with CYD dengue vaccine and classified as seronegative or undetermined at baseline in the Colombian study sites of CYD15, CYD13, CYD29, CYD64, or CYD65 trials
Sampling Method: Non-Probability Sample
Enrollment: 918 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-07-15 (Estimated)

PRIMARY OUTCOMES:
Type of access to care provided for participant with confirmed dengue | From Day 0 to end of participation (10 years after last dengue vaccination)
  Types of access are: urgent care/emergency room visit, hospitalization, medical care for suspected dengue case until dengue confirmation, diagnostic procedures and treatment, and medication
Virologically-confirmed dengue cases | From Day 0 to end of participation (10 years after last dengue vaccination)
  Dengue disease confirmed by NS1 Rapid Diagnostic Test in participant with suspected dengue
Suspected dengue case as per clinical diagnosis | From Day 0 to end of participation (10 years after last dengue vaccination)
  Suspected dengue is defined by high fever (40°C / 140 °F) and at least two of the following: nausea/vomiting, rash, aches and pain, tourniquet test positive, leukopenia, any warning sign

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Investigational site Colombia, Colombia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org